CLINICAL TRIAL: NCT02765698
Title: Efficacy of PET/MRI in Detecting Metastatic Disease in Endometrial Cancer
Status: Terminated | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Andrea Mariani, Professor of Obstetrics and Gynecology, Mayo Clinic
Other Study IDs: 15-004593
Record Dates: First submitted 2016-05-05; First posted 2016-05-09 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Endometrial Cancer
Keywords: Magnetic Resonance Imaging
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the ability of PET/MRI (Positron Emission Tomography/Magnetic Resonance Imaging) to give physicians preoperative information about specific sites in the body that the endometrial cancer may be present. If the PET/MRI is accurate and successful in providing this information, then women in the future may be able to have less extensive surgery for their endometrial cancer after evaluation with PET/MRI.

DETAILED DESCRIPTION:
PET/MRI has recently become available at the institution and reports of its sensitivity, specificity, NPV (Negative predictive value) , PPV (Positive predictive value), and accuracy in endometrial cancer are not found in the literature to date, to the best of the investigator's knowledge. The GE PET/MRI recently obtained here at Mayo, Rochester has the potential to improve the sensitivity of detection of metastatic disease, compared to other imaging modalities, because of its superior PET technology and updated Q Clear software. For these reasons it is reasonable to expect improved sensitivity to detect metastatic disease in endometrial cancer, possibly proving PET/MRI to be a superior modality for preoperative screening and potentially allowing for less morbid surgical management for patients with high risk endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven high-risk endometrial cancer (type 2 or grade 3 endometrioid histology)
* BMI of at least 18.5 kg/m2 and less than 35 kg/m2 or axial diameter less than 25 cm
* Patients who pass standard clinical MRI screening procedures
* Receiving preoperative clinical evaluation at Mayo Clinic, Rochester, MN
* Undergoing surgical staging and/or debulking at Mayo Clinic in Rochester, MN

Exclusion Criteria:

* Allergy to FDG or gadolinium
* Contraindication to MRI scanning (Extreme claustrophobia preventing PET/MRI completion, patients who are unable to lay quietly for an additional 60 minutes of imaging
* Known kidney disease or poor renal function
* Pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with biopsy-proven high risk (type 2 or grade 3 endometrioid histology) endometrial cancer undergoing debulking surgery.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2016-05; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Detection of distant metastasis of endometrial cancer by PET/MRI | one month
  Preoperative PET/MRI will be read by a radiologist and compared to final pathologic evaluation of metastatic specimens in high risk endometrial cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Mariani, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No